CLINICAL TRIAL: NCT05674435
Title: Clinical Utility of Neuromodulation on Tinnitus: A Systematic Review
Brief Title: Clinical Utility of Neuromodulation on Tinnitus
Status: Completed | Type: Observational
Sponsor: Hearing and Language Healthcare Center, China Medical University Hsinchu Hospital, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: IJS-D-22-01675
Record Dates: First submitted 2022-12-30; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present narrative review is to one of the first to critically evaluate the clinical effectiveness of neuromodulation as a therapeutic option for patients with tinnitus. Our method involves conducting a systemic review and the findings reported following PRISMA statement. Pubmed, Cochrane database and Google Scholar databases literature search was conducted for articles reporting the use of neuromodulatory interventions on tinnitus patients. Each article was evaluated using the Cochrane risk of bias tool.

ELIGIBILITY:
Inclusion Criteria:

* Tinnitus patients
* At least one of the neurofeedback methods
* Single and multi-center
* Randomized control trials and observational studies

Exclusion Criteria:

* Non-peer-reviewed papers, letters, editorials
* Not English language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tinnitus patients
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Tinnitus severity scores | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hearing and Language Healthcare Center, China Medical University Hsinchu Hospital, Taiwan, Hsinchu, Taiwan